CLINICAL TRIAL: NCT00995124
Title: A Randomised, Assessor Blind, Parallel Group, Comparative Trial of the Ovicidal Activity of Three Head Lice Products (NeutraLice Lotion®, NeutraLice Advance® and Moov Head Lice Solution®) After a Single Application
Brief Title: Trial of the Ovicidal Activity of Three Head Lice Products (NeutraLice Lotion®, NeutraLice Advance® and Moov Head Lice Solution®) After a Single Application
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Altman Biomedical Consulting Pty. Ltd. (Industry)
Responsible Party: Assoc. Prof. Stephen Barker, Parasitology Section, School of Chemistry & Molecular Biosciences, & UniQuest Pty Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEY/NL/003
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Head Lice
Keywords: ovicide; head lice infestation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NeutraLice Lotion (Experimental): Single application of head lice product.
  Interventions: Drug: NeutraLice Lotion
- NeutraLice Advance (Experimental): single application of head lice product
  Interventions: Drug: NeutraLice Advance Solution
- Moov Head Lice Solution (Active Comparator): Single application for head lice with 10 min application time.
  Interventions: Drug: Moov Head Lice Solution

INTERVENTIONS:
Drug: NeutraLice Lotion — Head lice topical application to be applied once for 10 minutes.
  Arms: NeutraLice Lotion
Drug: NeutraLice Advance Solution — head lice application to be applied once for 10 minutes
  Arms: NeutraLice Advance
Drug: Moov Head Lice Solution — Single application for head lice with 10 min application time.
  Arms: Moov Head Lice Solution

SUMMARY:
The purpose of this study is to compare the ovicidal activity of three head lice treatment products.

The study population will consist of Queensland primary school-aged children (Grades 1 - 7) who have at least 20 live eggs on the hair and who have not used any head lice product in the four weeks prior to the study.

Enrollment will continue to achieve 30 subjects in each treatment group (total of 90 subjects).

DETAILED DESCRIPTION:
Subjects will be examined for the presence of head louse eggs. Those subjects who have at least 20 live eggs will be randomised into one of 3 treatment groups: NeutraLice Lotion, NeutraLice Advance or Moov Head Lice Solution treatment groups.

Pre-treatment: 10 eggs will be removed from the head by cutting the single hair with the live egg attached, before the treatment.

Treatment: The subject will then receive a single treatment application according to manufacturers instructions. Then the treatment will be washed from the hair as per the manufacturer's instructions.

Post-treatment: At least 10 treated (live) eggs will be removed from the head by cutting the single hair with the egg attached, after the treatment.

All of the eggs will be held in an incubator for 14 days. The proportion of eggs which hatch after 14 days will be compared for the pre-treatment and post-treatment eggs. Demographic data will be collected for each subject (hair type, hair colour, hair length, subject age, subject sex) to investigate the affect of hair type on ovicidal efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female primary school-aged children.
* Presence of at least 20 live head lice eggs on the hair. The presence of live head lice eggs will be determined from a visual inspection of the hair.
* Parent / Guardian have given written informed consent to their child's participation in the trial.

Exclusion Criteria:

* History of allergies or adverse reactions to head lice products or the components of the specific products being tested.
* Treatment with any head lice product in the 4 weeks prior to participation in this trial.
* Treatment with hair dyes and bleaches within 4 weeks prior to participation in this trial.
* Presence of scalp disease(s).

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Ovicidal efficacy index (OEI) The proportion of treated eggs hatched in-vitro divided by the proportion of pre-treated eggs hatched in-vitro expressed as a percentage up to and including 14 days after collection and incubation. | ovicidal activity assessed after 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Barker, PhD, Principal Investigator — University of Queensland, Queensland, Australia
Locations (1):
- Assoc. Prof. Stephen Barker, Brisbane, New South Wales, Australia